CLINICAL TRIAL: NCT04542954
Title: Renal Dysfunction Among Patients With Severe Acute Respiratory Syndrome Coronavirus 2 (Covid-19) Patients: Kuwait Experience
Brief Title: Optimized Management of Covid-19 Positive Kidney Transplant Recipients: Single Center Experience From the Middle East
Acronym: OMC-KTR
Status: Completed | Type: Observational
Sponsor: Hamid Al-Essa Organ Transplant Center (Other Government)
Collaborators: Ministry of Health, Kuwait (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2020/1481
Record Dates: First submitted 2020-09-07; First posted 2020-09-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Covid19; Kidney Transplant Infection; Risk Factor, Cardiovascular; Immunosuppression; Outcome, Fatal; Graft Failure
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Optimized Management of Covid-19 Positive Kidney Transplant Recipients: Single Center Experience from the Middle East — Optimized Management of Covid-19 Positive Kidney Transplant Recipients: Single Center Experience from the Middle East

SUMMARY:
Methods: Out of 2000 kidney transplant recipients in our center in Kuwait, collecting data was started for all COVID-19-positive kidney transplant recipients till August 2020. Clinical features, management details and both patient and graft outcomes were reported.

DETAILED DESCRIPTION:
Before COVID-19 pandemic, nearly 2000 kidney transplant recipients were followed in our center in Kuwait. Data collection of such infected cases were started after diagnosing the 1st case during 1st week of March 2020. An ongoing study was performed that included 8 governmental acute care hospitals in Kuwait. All COVID-19-positive adult kidney transplant recipients with a functioning allograft who presented to the emergency department and were either discharged or hospitalized between March 1, 2020 and August 1, 2020 were included. Clinical features, management details and both patient and graft outcomes were reported. Data were collected from the electronic health record reporting database of both the mother transplant center and isolation hospitals.

Laboratory diagnosis:

COVID-19 positivity was defined as a positive result on real-time polymerase chain reaction (PCR) assay of nasopharyngeal swab specimens targeting the RNA-dependent RNA polymerase gene using amplification according to manufacturer's recommendation. Kidney transplant status was defined as an active International Statistical Classification of Diseases and Related Health Problems 10 code of T86.1, T86.10, T86.11, T86.12, T86.13, T86.19, or Z94.0. All electronic files were manually reviewed for demographics, history of recent exposure, immunosuppression changes, clinical signs and symptoms suggesting COVID-19, and laboratory findings with special stress on serum creatinine, liver function tests, D dimer, procalcitonin (PCT), C reactive protein and complete blood count. Acute kidney injury was graded according to Kidney Disease Improving Global Outcomes (KDIGO) criteria. AKI was staged for severity according to the following criteria: Stage 1 when creatinine was ranging between 1.5-<2 folds of basal; stage 2 if the creatinine was ranging between 2-<3folds and stage 3 if creatinine was more than 3 folds the basal. The study was approved by the ethical committee of ministry of health of Kuwait. Written informed consent was waived in light of the urgent need to collect data.

Radiological assessment:

The presence of a radiologic abnormality was determined on the basis of the documentation or description in medical charts of infected patients; if imaging scans were available, they were reviewed by attending physicians in respiratory medicine who extracted the data. If a major disagreement between two reviewers happened it was resolved by consultation with a third reviewer. The degree of severity of Covid-19 (severe vs. non-severe) at the time of admission will be defined using the American Thoracic Society guidelines for community-acquired pneumonia.7

Statistics:

Statistical analyses were conducted using SPSS version 20.0 (SPSS, Chicago, IL, USA). Qualitative data were presented as number and percent, and quantitative data were presented as means ± standard deviation and median. The t-test was used to compare means and standard deviations of the studied groups. Categorical data were compared using the chi-squared test. P values will be considered significant if < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* All renal transplant patients infected with COVID-19 during the period of 6 months from 3.2020 till the end of 8.2020

Exclusion Criteria:

* Pediatric patients

Age Groups: Child, Adult, Older Adult
Study Population: All Adult renal transplant patients infected with COVID-19 during the period of 6 months from 3.2020 till the end of 8.2020
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
patient outcome | 30 days
  living patients (1), dead patients(2) during the study period
Kidney graft outcome | 30 days
  functioning graft(1), failed graft(2) and impaired graft(3) at the end of the study

SECONDARY OUTCOMES:
risk factors for getting COVID19 infection | 30 days
  Diabetes(=!), IHD(=1), Hypertension(=1),pulmonary diseases(=1)

CONTACTS AND LOCATIONS:
Locations (1):
- OTC, MOH , Kuwait, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: No